CLINICAL TRIAL: NCT06674772
Title: Fenotipado Molecular De Pacientes Con Migraña Según Edad Y Sexo a Través De La Cuantificación De CGRP En Saliva Para Realizar Medicina De Precisión: Estudio FAST
Brief Title: Molecular Phenotyping of Migraine Patients According to Sex and Age Through CGRP Quantification
Acronym: FAST
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)350/2022
Record Dates: First submitted 2024-10-24; First posted 2024-11-05 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Headache (Migraine); Migraine; Migraine Headache; Migraine with Aura; Migraine Without Aura; Episodic Migraine; Chronic Migraine Headache; Chronic Migraine, Headache; Episodic Migraine Headache
Keywords: Migraine; CGRP; saliva
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood and saliva samples will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Migraine Patients: Patients, male and female, with Episodic migraine, all ages.
  Interventions: Diagnostic Test: Saliva test
- Control group: Male and female without migraine or headache
  Interventions: Diagnostic Test: Saliva test

INTERVENTIONS:
Diagnostic Test: Saliva test — Sampling of CGRP in saliva and DNA blood test and sex hormones blood test.
  Other Names: Blood test

SUMMARY:
Patients will be asked to visit the study center 2 times, the first time for clinical assessment and a second time for sample collection. Healthy controls will only be asked to visit the study center for sample collection. A sample of blood and saliva will be collected in order to measure CGRP levels and DNA and hormone testing.

DETAILED DESCRIPTION:
CGRP is a neuropeptide related to migraine pathophysiology, which can be found in human saliva in both patients and healthy controls. The differences in CGRP levels may help us explain the differences in the treatment response.

A sample of saliva will be collected in order to measure CGRP levels and a blood sample will be collected in order to conduct a DNA test and hormones test.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients according to ICHD-3 criteria
* Healthy controls paired to patient age and sex, without headache and without first degree family history of headache.

Exclusion Criteria:

* Presence of any major medical or neurological illness.
* Presence of any salivary gland malfunction.
* Abuse or dependence to tobacco, alcohol or any drug in the previous 12 months before the enrollment.
* Active migraine preventive treatment.
* Pregnant or breastfeeding female.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only cis-gender male and female will be included in the study due to hormone testing.
Study Population: Males and females otherwise healthy with episodic and chronic migraine in different age groups will be included in the study. Controls matching age and sex will be selected for the control groups.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
CGRP level | Through study completion, an average of 1 year
  Measure of CGRP in saliva
Hormone levels | Through study completion, an average of 1 year
  Blood test to quantify female hormones (FSH, LH, estradiol, progesterone, prolactin) and male hormones (testosterone) in all participants except for prepubertal children.
DNA test | Through study completion, an average of 1 year
  DNA testing for CGRP or its receptor related genes (CALCA, CALCB, CALCRL and RAMP1)

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided